CLINICAL TRIAL: NCT07151716
Title: Effect of Sedation With Dexmedetomidine-esketamine Combination on Delirium in Postoperative ICU Patients: a Randomized Controlled Pilot Trial
Brief Title: Sedation With Dexmedetomidine-esketamine Combination and Delirium in ICU Patients
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Peking University First Hospital (Other)
Responsible Party: Principal Investigator, Dong-Xin Wang, Professor and Chairman, Department of Anesthesiology, Peking University First Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2025R069
Record Dates: First submitted 2025-08-25; First posted 2025-09-03 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Older Patients; Postoperative Care; Intensive Care Unit; Dexmedetomidine; Esketamine; Delirium
Keywords: Older patients; Postoperative care; Intensive Care Unit; Dexmedetomidine; Esketamine; Delirium
MeSH Terms: conditions — Delirium | interventions — Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dexmedetomidine (Active Comparator): Sedation is provided with dexmedetomidine (4 μg/ml dexmedetomidine) for up to 7 days or until discharge from the ICU.
  Interventions: Drug: Dexmedetomidine
- Dexmedetomidine-esketamine combination (Experimental): Sedation is provided with dexmedetomidine-esketamine combination (2 μg/ml dexmedetomidine and 1 mg/ml esketamine) combination for up to 7 days or until discharge from the ICU.
  Interventions: Drug: Dexmedetomidine-esketamine combination

INTERVENTIONS:
Drug: Dexmedetomidine — For patients with endotracheal intubation, nighttime (20:00-06:00) sedation is initiated with 0.2 μg/kg/h dexmedetomidine and increased/decreased by 0.1 μg/kg/h dexmedetomidine every 15 min, until the Richmond Agitation-Sedation Scale (RASS) reaches -2 to -1, maximal infusion rate reaches 0.7 μg/kg/h dexmedetomidine, or adverse reactions occur. Daytime (06:00-20:00) sedation is provided as above when considered necessary, with a target RASS score of -2 to +1.
  For patients without endotracheal intubation, nighttime (20:00-06:00) sedation is initiated with 0.10 μg/kg/h dexmedetomidine and increased/decreased by 0.05 μg/kg/h dexmedetomidine every 15 min, until the RASS reaches -1, maximal infusion rate reaches 0.2 μg/kg/h dexmedetomidine, or adverse reactions occur. Daytime (06:00-20:00) sedation is typically not provided.
  Other Names: Sedation with dexmedetomidine
  Arms: Dexmedetomidine
Drug: Dexmedetomidine-esketamine combination — For patients with endotracheal intubation, nighttime (20:00-06:00) sedation is initiated with 0.1 μg/kg/h dexmedetomidine and 0.05 mg/kg/h esketamine, increased/decreased by 0.05 μg/kg/h dexmedetomidine and 0.025 mg/kg/h esketamine every 15 min, until the RASS reaches -2 to -1, maximal infusion rate reaches 0.35 μg/kg/h dexmedetomidine and 0.175 mg/kg/h esketamine, or adverse reactions occur. Daytime (06:00-20:00) sedation is provided as above when considered necessary, with a target RASS score of -2 to +1.
  For patients without endotracheal intubation, nighttime (20:00-06:00) sedation is initiated with 0.05 μg/kg/h dexmedetomidine and 0.025 mg/kg/h esketamine, and increased/decreased by 0.025 μg/kg/h dexmedetomidine and 0.0125 mg/kg/h esketamine every 15 min, until the RASS reaches -1, maximal infusion rate reaches 0.1 μg/kg/h dexmedetomidine and 0.05 mg/kg/h esketamine, or adverse reactions occur. Daytime (06:00-20:00) sedation is typically not provided.
  Other Names: Sedation with dexmedetomidine-esketamine combination
  Arms: Dexmedetomidine-esketamine combination

SUMMARY:
Patients in the intensive care unit (ICU) often develop anxiety and agitation, sleep disturbances, and delirium. Delirium occurrence is associated with worse early and long-term outcomes. Dexmedetomidine and ketamine are recommended for sedation and analgesia in postoperative ICU patients, but each may induce side effects. The sedative effects of dexmedetomidine can help mitigate the neuropsychiatric side effects of esketamine. Recent studies showed that dexmedetomidine-esketamine combination improved analgesia and sleep quality without increasing side effects. This trial is designed to test the hypothesis that dexmedetomidine-esketamine combination for sedation and analgesia in postoperative ICU patients may reduce delirium.

DETAILED DESCRIPTION:
An estimated 300 million surgical procedures are performed globally each year. Patients who have complex conditions and an elevated risk of postoperative complications frequently require admission to the intensive care unit (ICU). Among these, a subset are admitted to ICU with an endotracheal tube and continue to receive mechanical ventilation. Sleep disturbances are highly prevalent in ICU patients due to environmental factors, underlying diseases, therapeutic interventions, and pain-related stimuli.

Mechanical ventilation, painful stimulation, and sleep disturbances are important risk factors of delirium in ICU patients. Delirium is an acutely occurred brain dysfunction symdrome characteristized with fluctuating disturbances in attention, cognition, and consciousness, and is reported to occur in up to 80% of ICU patients with mechanical ventilation. Delirium occurrence is associated with worse outcomes, including prolonged mechanical ventilation, extended ICU and hospital stays, increased healthcare burden and costs, and elevated mortality risk, as well as long-term sequelae including cognitive decline, reduced quality of life, and decreased survival.

Dexmedetomidine is a highly selective α2-adrenergic receptor agonist with sedative, analgesic, and anxiolytic effects. It exerts effects by activating the endogenous sleep-promoting pathways, inducing a state like non-rapid eye movement sleep. Ketamine is a non-competitive N-methyl-D-aspartate (NMDA) receptor antagonist. Esketamine, a more potent enantiomer of ketamine, has a higher affinity for the NMDA receptor and is approximately twice as potent as ketamine. Both dexmedetomidine and ketamine are recommended for sedation and analgesia in postoperative ICU patients. However, sedative dose dexmedetomidine is associated with bradycardia and hypotension. Even low-dose esketamine can induce neuropsychiatric side effects such as dissociation, hallucinations, and nightmares.

The sedative effects of dexmedetomidine can help mitigate the neuropsychiatric side effects of esketamine. Recent studies showed that low-dose dexmedetomidine-esketamine combination improved analgesia and sleep quality without increasing side effects. It is hypothesized that dexmedetomidine-esketamine combination for sedation and analgesia in postoperative ICU patients may reduce delirium.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 60 years or older;
2. Admitted to the intensive care unit (ICU) after surgery;
3. Expected to stay in the ICU for at least one night.

Exclusion Criteria:

1. History of schizophrenia, epilepsy, Parkinson's disease, or myasthenia gravis;
2. Presence of preoperative delirium, or inability to communicate due to coma, severe dementia, or language barrier;
3. Previously diagnosed obstructive sleep apnea, judged to be at high risk of moderate-to-severe obstructive sleep apnea according to the STOP-Bang questionnaire, or have a body mass index >30 kg/m²;
4. Preoperative left ventricular ejection fraction <30%, sick sinus syndrome, severe sinus bradycardia (heart rate <50 bpm), second-degree or higher atrioventricular block without a pacemaker, or systolic blood pressure <90 mmHg despite use of vasopressors;
5. Comorbid with hyperthyroidism or pheochromocytoma;
6. Severe liver dysfunction (Child-Pugh Class C), severe renal dysfunction (requiring dialysis), or expected survival ≤24 hours;
7. After traumatic brain injury or neurosurgery;
8. Allergy to dexmedetomidine and/or esketamine;
9. Other conditions that are considered unsuitable for study participation.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-10-21 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Incidence of delirium within 7 days | Up to 7 days after surgery
  Delirium will be assessed twice daily (8:00-10:00, 18:00-20:00) for 7 days or until hospital discharge. Patients with endotracheal intubation will be assessed with the Confusion Assessment Method for the Intensive Care Unit (CAM-ICU). Patients without endotracheal intubation will be assessed with the 3-Minute Diagnostic Assessment for Delirium using the Confusion Assessment Method (3D-CAM). Positive result of delirium assessments at any timepoint is defined as occurrence of delirium.

SECONDARY OUTCOMES:
Total sleep time (TST) on the first postoperative night | From 20:00 on the night of surgery to 06:00 the next morning
  Total sleep time will be monitored using an actigraphy device.
Postoperative pain score within 7 days | Up to 7 days after surgery
  Pain intensity will be assessed twice daily (8:00-10:00, 18:00-20:00) for 7 days or until hospital discharge, using the 11-point Numeric Rating Scale (NRS; 0 = no pain, 10 = worst pain) or the Behavioral Pain Scale (BPS; range 4-16, with higher scores indicating more severe pain; for patients with deep sedation).
Postoperative subjective sleep quality within 7 days | Up to 7 days after surgery
  Subjective sleep quality will be assessed once daily (08:00-10:00) for 7 days or until hospital discharge, using an 11-point Numeric Rating Scale (0 = best sleep, 10 = worst sleep)
Length of stay in the ICU | Up to 30 days after surgery
  Length of stay in the ICU

OTHER OUTCOMES:
Length of stay in hospital after surgery | Up to 30 days after surgery
  Length of stay in hospital after surgery
Incidence of major complications within 30 days | Up to 30 days after surgery
  Major complications are defined as new-onset medical conditions other than delirium that are deemed harmful and require therapeutic intervention, that is grade II or higher on the Clavien-Dindo classification.
Incidence of cognitive dysfunction at 30 days | At 30 days after surgery
  Cognitive function is assessed with the Montreal Cognitive Assessment-telephone version (T-MoCA; score ranges from 0 to 22, with higher score indicating better cognitive function). A decline of 1 standard deviation (SD) or more from baseline is defined as having cognitive dysfunction.
Concentration of amyloid-β peptide 42 (Aβ42) in plasma (part of patients) | On the morning of the 1st postoperative day
  Concentration of amyloid-β peptide 42 (Aβ42) in plasma on the morning of the 1st postoperative day
Concentration of phosphorylated tau at threonine 217 (Tau-PT217) in plasma (part of patients) | On the morning of the 1st postoperative day
  Concentration of phosphorylated tau at threonine 217 (Tau-PT217) in plasma on the morning of the 1st postoperative day
Concentration of phosphorylated tau at threonine 181 (Tau-PT181) in plasma (part of patients) | On the morning of the 1st postoperative day
  Concentration of phosphorylated tau at threonine 181 (Tau-PT181) in plasma on the morning of the 1st postoperative day
Concentration of S100 calcium binding protein B (S100B) in plasma (part of patients) | On the morning of the 1st postoperative day
  Concentration of S100 calcium binding protein B (S100B) in plasma on the morning of the 1st postoperative day
Concentration of glial fibrillary acidic protein (GFAP) in plasma (part of patients) | On the morning of the 1st postoperative day
  Concentration of glial fibrillary acidic protein (GFAP) in plasma on the morning of the 1st postoperative day
Concentration of interleukin-1 beta (IL-1β) in plasma (part of patients) | On the morning of the 1st postoperative day
  Concentration of interleukin-1 beta (IL-1β) in plasma on the morning of the 1st postoperative day
Concentration of interleukin-6 (IL-6) in plasma (part of patients) | On the morning of the 1st postoperative day
  Concentration of interleukin-6 (IL-6) in plasma on the morning of the 1st postoperative day
Concentration of interleukin-10 (IL-10) in plasma (part of patients) | On the morning of the 1st postoperative day
  Concentration of interleukin-10 (IL-10) in plasma on the morning of the 1st postoperative day
Concentration of tumor necrosis factor-alpha (TNF-α) in plasma (part of patients) | On the morning of the 1st postoperative day
  Concentration of tumor necrosis factor-alpha (TNF-α) in plasma on the morning of the 1st postoperative day

CONTACTS AND LOCATIONS:
Overall Officials: Dong-Xin Wang, MD, PhD, Principal Investigator — Peking University First Hospital
Locations (1):
- Peking University First Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wang S, Yu X, Cheng L, Ren W, Wen G, Wu X, Lou H, Ren X, Lu L, Hermenean A, Yao J, Li B, Lu Y, Wu X. Dexmedetomidine improves the circulatory dysfunction of the glymphatic system induced by sevoflurane through the PI3K/AKT/DeltaFosB/AQP4 pathway in young mice. Cell Death Dis. 2024 Jun 25;15(6):448. doi: 10.1038/s41419-024-06845-w. PMID 38918408
- [Background] Dong R, Liu W, Han Y, Wang Z, Jiang L, Wang L, Gu X. Influencing factors of glymphatic system during perioperative period. Front Neurosci. 2024 Sep 12;18:1428085. doi: 10.3389/fnins.2024.1428085. eCollection 2024. PMID 39328423
- [Background] Lewis K, Balas MC, Stollings JL, McNett M, Girard TD, Chanques G, Kho ME, Pandharipande PP, Weinhouse GL, Brummel NE, Chlan LL, Cordoza M, Duby JJ, Gelinas C, Hall-Melnychuk EL, Krupp A, Louzon PR, Tate JA, Young B, Jennings R, Hines A, Ross C, Carayannopoulos KL, Aldrich JM. A Focused Update to the Clinical Practice Guidelines for the Prevention and Management of Pain, Anxiety, Agitation/Sedation, Delirium, Immobility, and Sleep Disruption in Adult Patients in the ICU. Crit Care Med. 2025 Mar 1;53(3):e711-e727. doi: 10.1097/CCM.0000000000006574. Epub 2025 Feb 21. PMID 39982143
- [Background] Alexopoulou C, Kondili E, Diamantaki E, Psarologakis C, Kokkini S, Bolaki M, Georgopoulos D. Effects of dexmedetomidine on sleep quality in critically ill patients: a pilot study. Anesthesiology. 2014 Oct;121(4):801-7. doi: 10.1097/ALN.0000000000000361. PMID 24988068
- [Background] Nelson LE, Lu J, Guo T, Saper CB, Franks NP, Maze M. The alpha2-adrenoceptor agonist dexmedetomidine converges on an endogenous sleep-promoting pathway to exert its sedative effects. Anesthesiology. 2003 Feb;98(2):428-36. doi: 10.1097/00000542-200302000-00024. PMID 12552203
- [Background] Weerink MAS, Struys MMRF, Hannivoort LN, Barends CRM, Absalom AR, Colin P. Clinical Pharmacokinetics and Pharmacodynamics of Dexmedetomidine. Clin Pharmacokinet. 2017 Aug;56(8):893-913. doi: 10.1007/s40262-017-0507-7. PMID 28105598
- [Background] Kanji S, Mera A, Hutton B, Burry L, Rosenberg E, MacDonald E, Luks V. Pharmacological interventions to improve sleep in hospitalised adults: a systematic review. BMJ Open. 2016 Jul 29;6(7):e012108. doi: 10.1136/bmjopen-2016-012108. PMID 27473952
- [Background] Weinhouse GL, Watson PL. Sedation and sleep disturbances in the ICU. Crit Care Clin. 2009 Jul;25(3):539-49, ix. doi: 10.1016/j.ccc.2009.04.003. PMID 19576529
- [Background] Trompeo AC, Vidi Y, Locane MD, Braghiroli A, Mascia L, Bosma K, Ranieri VM. Sleep disturbances in the critically ill patients: role of delirium and sedative agents. Minerva Anestesiol. 2011 Jun;77(6):604-12. PMID 21617624
- [Background] Mehta S, Cook D, Devlin JW, Skrobik Y, Meade M, Fergusson D, Herridge M, Steinberg M, Granton J, Ferguson N, Tanios M, Dodek P, Fowler R, Burns K, Jacka M, Olafson K, Mallick R, Reynolds S, Keenan S, Burry L; SLEAP Investigators; Canadian Critical Care Trials Group. Prevalence, risk factors, and outcomes of delirium in mechanically ventilated adults. Crit Care Med. 2015 Mar;43(3):557-66. doi: 10.1097/CCM.0000000000000727. PMID 25493968
- [Background] Ely EW, Inouye SK, Bernard GR, Gordon S, Francis J, May L, Truman B, Speroff T, Gautam S, Margolin R, Hart RP, Dittus R. Delirium in mechanically ventilated patients: validity and reliability of the confusion assessment method for the intensive care unit (CAM-ICU). JAMA. 2001 Dec 5;286(21):2703-10. doi: 10.1001/jama.286.21.2703. PMID 11730446
- [Background] Krewulak KD, Stelfox HT, Leigh JP, Ely EW, Fiest KM. Incidence and Prevalence of Delirium Subtypes in an Adult ICU: A Systematic Review and Meta-Analysis. Crit Care Med. 2018 Dec;46(12):2029-2035. doi: 10.1097/CCM.0000000000003402. PMID 30234569
- [Background] Mattimore D, Fischl A, Christophides A, Cuenca J, Davidson S, Jin Z, Bergese S. Delirium after Cardiac Surgery-A Narrative Review. Brain Sci. 2023 Dec 7;13(12):1682. doi: 10.3390/brainsci13121682. PMID 38137130
- [Background] Igwe EO, Nealon J, O'Shaughnessy P, Bowden A, Chang HR, Ho MH, Montayre J, Montgomery A, Rolls K, Chou KR, Chen KH, Traynor V, Smerdely P. Incidence of postoperative delirium in older adults undergoing surgical procedures: A systematic literature review and meta-analysis. Worldviews Evid Based Nurs. 2023 Jun;20(3):220-237. doi: 10.1111/wvn.12649. Epub 2023 May 2. PMID 37128953
- [Background] Wilson JE, Mart MF, Cunningham C, Shehabi Y, Girard TD, MacLullich AMJ, Slooter AJC, Ely EW. Delirium. Nat Rev Dis Primers. 2020 Nov 12;6(1):90. doi: 10.1038/s41572-020-00223-4. PMID 33184265
- [Background] Slatore CG, Goy ER, O'hearn DJ, Boudreau EA, O'Malley JP, Peters D, Ganzini L. Sleep quality and its association with delirium among veterans enrolled in hospice. Am J Geriatr Psychiatry. 2012 Apr;20(4):317-26. doi: 10.1097/JGP.0b013e3182487680. PMID 22367162
- [Background] Van Rompaey B, Elseviers MM, Schuurmans MJ, Shortridge-Baggett LM, Truijen S, Bossaert L. Risk factors for delirium in intensive care patients: a prospective cohort study. Crit Care. 2009;13(3):R77. doi: 10.1186/cc7892. Epub 2009 May 20. PMID 19457226
- [Background] Fong HK, Sands LP, Leung JM. The role of postoperative analgesia in delirium and cognitive decline in elderly patients: a systematic review. Anesth Analg. 2006 Apr;102(4):1255-66. doi: 10.1213/01.ane.0000198602.29716.53. PMID 16551934
- [Background] Miner SE, Pahal D, Nichols L, Darwood A, Nield LE, Wulffhart Z. Sleep Disruption is Associated with Increased Ventricular Ectopy and Cardiac Arrest in Hospitalized Adults. Sleep. 2016 Apr 1;39(4):927-35. doi: 10.5665/sleep.5656. PMID 26715226
- [Background] Tobaldini E, Fiorelli EM, Solbiati M, Costantino G, Nobili L, Montano N. Short sleep duration and cardiometabolic risk: from pathophysiology to clinical evidence. Nat Rev Cardiol. 2019 Apr;16(4):213-224. doi: 10.1038/s41569-018-0109-6. PMID 30410106
- [Background] Fernandes NM, Nield LE, Popel N, Cantor WJ, Plante S, Goldman L, Prabhakar M, Manlhiot C, McCrindle BW, Miner SE. Symptoms of disturbed sleep predict major adverse cardiac events after percutaneous coronary intervention. Can J Cardiol. 2014 Jan;30(1):118-24. doi: 10.1016/j.cjca.2013.07.009. Epub 2013 Oct 16. PMID 24140074
- [Background] Sharma V, Rao V, Manlhiot C, Boruvka A, Fremes S, Wasowicz M. A derived and validated score to predict prolonged mechanical ventilation in patients undergoing cardiac surgery. J Thorac Cardiovasc Surg. 2017 Jan;153(1):108-115. doi: 10.1016/j.jtcvs.2016.08.020. Epub 2016 Aug 29. PMID 27665221
- [Background] Tate JA, Devito Dabbs A, Hoffman LA, Milbrandt E, Happ MB. Anxiety and agitation in mechanically ventilated patients. Qual Health Res. 2012 Feb;22(2):157-73. doi: 10.1177/1049732311421616. Epub 2011 Sep 9. PMID 21908706
- [Background] May AD, Parker AM, Caldwell ES, Hough CL, Jutte JE, Gonzalez MS, Needham DM, Hosey MM. Provider-Documented Anxiety in the ICU: Prevalence, Risk Factors, and Associated Patient Outcomes. J Intensive Care Med. 2021 Dec;36(12):1424-1430. doi: 10.1177/0885066620956564. Epub 2020 Oct 9. PMID 33034254
- [Background] Honarmand K, Rafay H, Le J, Mohan S, Rochwerg B, Devlin JW, Skrobik Y, Weinhouse GL, Drouot X, Watson PL, McKinley S, Bosma KJ. A Systematic Review of Risk Factors for Sleep Disruption in Critically Ill Adults. Crit Care Med. 2020 Jul;48(7):1066-1074. doi: 10.1097/CCM.0000000000004405. PMID 32433122
- [Background] Hardin KA, Seyal M, Stewart T, Bonekat HW. Sleep in critically ill chemically paralyzed patients requiring mechanical ventilation. Chest. 2006 Jun;129(6):1468-77. doi: 10.1378/chest.129.6.1468. PMID 16778263
- [Background] Cooper AB, Thornley KS, Young GB, Slutsky AS, Stewart TE, Hanly PJ. Sleep in critically ill patients requiring mechanical ventilation. Chest. 2000 Mar;117(3):809-18. doi: 10.1378/chest.117.3.809. PMID 10713011
- [Background] Zampieri FG, Lone NI, Bagshaw SM. Admission to intensive care unit after major surgery. Intensive Care Med. 2023 May;49(5):575-578. doi: 10.1007/s00134-023-07026-7. Epub 2023 Mar 22. No abstract available. PMID 36947198
- [Background] Ohbe H, Matsui H, Kumazawa R, Yasunaga H. Postoperative ICU admission following major elective surgery: A nationwide inpatient database study. Eur J Anaesthesiol. 2022 May 1;39(5):436-444. doi: 10.1097/EJA.0000000000001612. Epub 2021 Oct 11. PMID 34636358
- [Background] Weiser TG, Haynes AB, Molina G, Lipsitz SR, Esquivel MM, Uribe-Leitz T, Fu R, Azad T, Chao TE, Berry WR, Gawande AA. Estimate of the global volume of surgery in 2012: an assessment supporting improved health outcomes. Lancet. 2015 Apr 27;385 Suppl 2:S11. doi: 10.1016/S0140-6736(15)60806-6. Epub 2015 Apr 26. PMID 26313057